CLINICAL TRIAL: NCT07169487
Title: Exploration of Efficacy and Safety of Adjunctive Methylene Blue in the Treatment of Immunotherapy-related CRS and ICANS: A Prospective, Single-arm, Phase I Clinical Study
Brief Title: Adjunctive Methylene Blue for Immunotherapy-related CRS and ICANS: Phase I Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025072
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cytokine Release Syndrome; ICANS
Keywords: Methylene Blue; Cytokine Release Syndrome; Immune Effector Cell-Associated Neurotoxicity Syndrome; CAR-T Cell Therapy; Immunotherapy-Related Toxicity
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjunctive Methylene Blue Dose-Escalation in Immunotherapy-related CRS and ICANS (Experimental): To evaluate the efficacy and safety of adjunctive methylene blue in the treatment of immunotherapy-related cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) in patients receiving CAR-T or bispecific antibody therapy, using a 3+3 dose-escalation Phase I design.
  Interventions: Drug: Methylene Blue

INTERVENTIONS:
Drug: Methylene Blue — Intravenous infusion of methylene blue once daily for 3-5 consecutive days at doses of 1 mg/kg, 2 mg/kg, or 3 mg/kg, administered over 20 minutes, following CAR-T or bispecific antibody infusion in patients who develop Grade ≥1 CRS or ICANS.

SUMMARY:
This Phase I, prospective, single-arm clinical study aims to evaluate the efficacy and safety of adjunctive methylene blue (MB) in patients experiencing cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS) following CAR-T cell therapy or bispecific antibody treatment. Preclinical studies demonstrated that MB alleviates CRS/ICANS-related symptoms, preserves the antitumor function of T cells, and modulates neuroinflammation without compromising immune efficacy. The study will employ a 3+3 dose-escalation design with three MB dosing cohorts, with treatment administered intravenously for 3-5 consecutive days. Vital signs, laboratory markers, and neurological status will be closely monitored, and concomitant standard supportive therapies will be permitted.

DETAILED DESCRIPTION:
Methylene blue (MB), originally approved for methemoglobinemia, has demonstrated hemodynamic and neuroprotective effects. Preclinical data indicate that MB alleviates CRS/ICANS symptoms, protects blood-brain barrier integrity, limits microglial overactivation, and preserves T-cell antitumor function.

This Phase I, prospective, single-arm clinical trial will investigate MB as an adjunctive therapy for immunotherapy-related CRS and ICANS. Eligible patients are those receiving CAR-T cells or bispecific antibodies who subsequently develop Grade ≥1 CRS or ICANS, as defined by ASTCT 2019 criteria. Participants will be enrolled in a 3+3 dose-escalation schema with the following cohorts:

Cohort 1: 1 mg/kg once daily, intravenous infusion over 20 minutes Cohort 2: 2 mg/kg once daily, intravenous infusion over 20 minutes Cohort 3: 3 mg/kg once daily, intravenous infusion over 20 minutes Treatment will be administered for 3-5 consecutive days. Patients will undergo continuous assessment of vital signs (temperature, blood pressure, oxygen saturation), laboratory biomarkers (CRP, ferritin, cytokines), and neurotoxicity grading throughout therapy. Dosing adjustments will be based on real-time safety and efficacy evaluations.

Concomitant standard-of-care supportive interventions will be allowed, including tocilizumab (maximum of two doses), dexamethasone, ruxolitinib, cetuximab, and other symptomatic treatments. This trial seeks to establish the safety profile and preliminary efficacy of MB in mitigating immune therapy-related toxicities, potentially offering a novel strategy to improve the tolerability and safety of CAR-T and bispecific antibody therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hematologic malignancies based on cytomorphology and immunophenotyping; age ≥18 years.
2. Received immunotherapy (e.g., CAR-T cells, bispecific antibodies) and developed CRS or ICANS of ASTCT Grade ≥1.
3. Estimated life expectancy ≥3 months.
4. Male and female participants of childbearing potential agree to use effective contraception.
5. Left ventricular ejection fraction (LVEF) >45% by echocardiography.
6. Ability to understand and sign informed consent and willingness to comply with study requirements.

Exclusion Criteria:

1. Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
2. Known allergy to methylene blue.
3. Pregnant or breastfeeding women.
4. Known HIV seropositivity. HIV testing may be required according to local laws or regulations.
5. History of clinically significant ventricular arrhythmia, unexplained syncope (not vasovagal), sinoatrial block, or higher-degree atrioventricular (AV) block with chronic bradycardia (unless a permanent pacemaker is implanted).
6. Psychiatric disorders that may interfere with completion of treatment or informed consent.
7. Any other condition deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2030-06-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of methylene blue-related serious adverse events (SAEs) | Up to Day 35 after initiation of methylene blue treatment
  The proportion of participants who experience methylene blue-related serious adverse events (SAEs), categorized by type, assessed according to NCI CTCAE v5.0 criteria. SAEs will be judged by the investigator to be related to methylene blue administration.
Impact of Methylene Blue on CAR-T/T Cell Expansion in Peripheral Blood | Up to Day 35 after initiation of methylene blue treatment
  Evaluation of CAR-T or T cell expansion in peripheral blood following methylene blue treatment, assessed by flow cytometry.
Impact of Methylene Blue on CAR-T/T Cell Therapy Efficacy | Baseline to Day 35 post-treatment initiation
  Proportion of participants achieving complete remission (CR), partial remission (PR), stable disease (SD), or experiencing relapse/progression, assessed according to immunotherapy response criteria (see Study Protocol for full criteria).

SECONDARY OUTCOMES:
Incidence of Grade ≥3 CRS and ICANS | Up to Day 35 after initiation of methylene blue treatment
  Proportion of participants who develop Grade 3 or higher cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS), assessed according to ASTCT 2019 grading criteria.
Duration of CRS and ICANS | Up to Day 35 after initiation of methylene blue treatment
  The total duration (in days) of CRS and ICANS from onset until resolution to Grade 0, according to ASTCT 2019 criteria.
Duration of corticosteroid use | Up to Day 35 after initiation of methylene blue treatment
  Total duration (in days) of systemic corticosteroid administration for the management of CRS and/or ICANS after initiation of methylene blue treatment.
Proportion of Participants Requiring Vasopressors | Up to Day 35 after initiation of methylene blue treatment
  Percentage of participants who required vasopressor therapy at any time after initiation of methylene blue treatment.
Duration of Vasopressor Therapy | Up to Day 35 after initiation of methylene blue treatment
  Total number of days participants received vasopressor therapy after initiation of methylene blue treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China